CLINICAL TRIAL: NCT02541994
Title: The Potential Value of Axial Length and Central Corneal Thickness in the Assessment for Risk of Permanent Optic Nerve Damage and Visual Field Loss in Benign Intracranial Hypertension
Brief Title: Axial Length and Central Corneal Thickness in Benign Intracranial Hypertension
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Disparate corneal thickness readings from two measurement techniques employed.
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Andrew Lawton, MD, Physician, Ochsner Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2015.002.A
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Results first posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Benign Intracranial Hypertension
MeSH Terms: conditions — Pseudotumor Cerebri

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound Testing (Other): Single arm with all patients getting measurements of axial length and central corneal thickness.
  Interventions: Device: Pachette3; Device: Lenstar-Think

INTERVENTIONS:
Device: Pachette3 — Central corneal thickness will be measured with an ultrasound probe. This test will be performed while the corneas are anesthetized. This test will be performed as part of a standard, comprehensive dilated eye examination with optical coherence tomography and visual field testing as the regular care for benign intracranial hypertension.
  Other Names: Serial Number 2008-1206; Model DGH555
Device: Lenstar-Think — Axial length will be measured with an ultrasound probe. This test will be performed while the corneas are anesthetized. This test will be performed as part of a standard, comprehensive dilated eye examination with optical coherence tomography and visual field testing as the regular care for benign intracranial hypertension.
  Other Names: Model LS900; Serial Number 02114

SUMMARY:
Patients in for treatment of benign intracranial hypertension will undergo two tests that are not routinely performed for these patients: central corneal thickness and axial length of the eye. The data obtained from these measurements will be assessed to see if the correlate with aspects of vision loss including visual acuity, visual field status, optical coherence tomography (OCT) results, and fundus photographs.

DETAILED DESCRIPTION:
Patients with benign intracranial hypertension would be identified at diagnosis from the general ophthalmic and neurologic patient population in the Ochsner Health System. All would have a baseline eye examination with visual field and optical coherence tomography (OCT) testing, a standard step in managing any patient with this condition. Two measurements would be taken at minimal risk to the patient that they would not normally have done at the baseline exam: central corneal thickness and axial length. These procedures are routinely done on patients with glaucoma, corneal disease, and cataracts without a significant risk of injury. The theoretical risks with central corneal thickness and axial length measurements by A-scan ultrasonography are related to the small risk for transmission of infection or corneal abrasion due to a probe touching the cornea. These tests would be performed at no charge to the patient and would not significantly increase the time of the ocular examination. Patients would have neuro-imaging studies and lumbar puncture to confirm the diagnosis of benign intracranial hypertension as standard parts of the work up for the condition independent of the research study. The authors will statistically analyze the standard measures of visual field function and health of the nerve fiber layer by OCT to see if any or all of the proposed risk factors correlates with deterioration of visual function. Data would continue to be collected at follow up visits related to visual fields and OCT as would normally be performed on standard visits for this condition. The measurements of central corneal thickness and axial length would be performed solely at the time of enrollment in the study since these measurements do not change over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have benign intracranial hypertension.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Lawton, MD, Principal Investigator — Ochsner Health Services

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Testing
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound Testing
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (7.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Axial Length
Description: The length of the eye will be measured with ultrasound.
Time Frame: Single measurement during ultrasound procedure on the day of enrollment in the study on average of 5 minutes.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Ultrasound Testing
Number analyzed (Participants) | 5
millimeter | 23.67 (1.31)

2. Secondary Outcome: Central Corneal Thickness
Description: The thickness of the cornea will be measured with ultrasound.
Time Frame: Single measurement during ultrasound procedure at the time of enrollment in the study on average of 5 minutes.
Population: 10 eyes
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Ultrasound Testing
Number analyzed (Participants) | 5
Microns | 556.3 (26.9)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ultrasound Testing
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No